CLINICAL TRIAL: NCT01090050
Title: Treximet in the Treatment of Chronic Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cady, Roger, M.D. (Individual)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112839
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Results first posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Migraine
Keywords: Chronic Migraine; Migraine; Treximet; naproxen; sumatriptan
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan; Naproxen; sumatriptan-naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sumatriptan/Naproxen Sodium (Active Comparator): In Treatment Period Month 1: Subjects randomized to Sumatriptan/Naproxen Sodium will treat daily with 1 tablet Sumatriptan 85mg / Naproxen Sodium 500mg per day x 30 days. Subjects will be provided with 30 tablets of Sumatriptan/Naproxen Sodium for rescue. In Treatment Period Months 2 and 3: Subjects randomized to Sumatriptan/Naproxen Sodium will be provided with 14 tablets of Sumatriptan/Naproxen Sodium to treat on 14 or fewer days per month. Subjects will be provided with 14 tablets of Sumatriptan/Naproxen Sodium per month for rescue.
  Interventions: Drug: Sumatriptan/Naproxen Sodium
- Naproxen Sodium (Active Comparator): In Treatment Period Month 1: Subjects randomized to Naproxen Sodium will treat daily with 1 tablet Naproxen Sodium 500mg per day x 30 days. Subjects will be provided with 30 tablets of Naproxen Sodium for rescue. In Treatment Period Months 2 and 3: Subjects randomized to Naproxen Sodium will be provided with 14 tablets of Naproxen Sodium to treat on 14 or fewer days per month. Subjects will be provided with 14 tablets of Naproxen Sodium per month for rescue.
  Interventions: Drug: Naproxen Sodium

INTERVENTIONS:
Drug: Sumatriptan/Naproxen Sodium — Each tablet of Sumatriptan/Naproxen Sodium for oral administration contains sumatriptan 85mg / naproxen sodium 500mg. Study medication is to be administered 1 tablet per day x 30 days in Treatment Period Month 1. Study medication may be administered on up to 14 days per month in Treatment Period Months 2 and 3.
  Other Names: Treximet
  Arms: Sumatriptan/Naproxen Sodium
Drug: Naproxen Sodium — Each tablet of Naproxen Sodium for oral administration is provided in 500mg tablet. Study medication is to be administered 1 tablet per day x 30 days in Treatment Period Month 1. Study medication may be administered on up to 14 days per month in Treatment Period Months 2 and 3.
  Arms: Naproxen Sodium

SUMMARY:
This study is being conducted to evaluate the hypothesis that use of Treximet in patients with chronic migraine, when used on a short term daily basis and as rescue for break through attacks, will reduce migraine frequency and impact.

DETAILED DESCRIPTION:
One investigative center will enroll 40 subjects in the US.

At Visit 1, following informed consent, a medical, migraine, and medication history will be collected and a physical and neurological exam with vital signs will be performed. A 12-lead ECG will be completed. Eligible subjects will complete a 1-month Baseline Period and treat migraine with their current preferred treatment of choice. Throughout the study, subjects will complete daily Headache Diaries reporting headache severity and associated symptoms with use of study medication in each 30-day period.

At Visit 2, subjects continuing to meet eligibility criteria will be randomized 1:1 to Treximet or naproxen and provided with medication to treat daily for 30 days. At Visits 3 and 4 subjects will be provided with study medication to treat on 14 or fewer days per month. Subjects will be encouraged to treat their migraine attacks within 1 hour of onset of headache pain and while the pain is still mild. Adverse events will be collected beginning from the first dose of study medication. Subjects exit the study at Visit 5 after a 3-month Treatment Period.

The study provides opportunity to evaluate the usefulness of patient education with a 15-minute digital versatile disc (DVD) concerning the processes of headache evolution and lifestyle changes for better headache management. At Visit 2, subjects will view the DVD in-clinic with a copy provided for at-home viewing. Subjects will complete a Lifestyle Choices for Better Migraine Management Questionnaire at each visit and receive 3 copies to be completed weekly and returned at the following visit.

The Migraine Disability Assessment questionnaire (MIDAS) will be completed at Visits 2 and 5 to determine the level of pain and disability caused by headache.

ELIGIBILITY:
Inclusion Criteria:

Subject

* Is male or female, in otherwise good health, 18 to 65 years of age.
* Has history of chronic migraine (with or without aura) according to the criteria proposed by the Headache Classification Committee of the International Headache Society for at least 3 months prior to enrollment.
* Has onset of migraine before age 50.
* Is able to differentiate migraine from any other headache they may experience (e.g., tension-type headache).
* Has stable history of headache for at least 3 months prior to screening.
* Is not currently taking a migraine preventive or has been taking preventive for at least 30 days prior to screening and agrees to not start, stop, or change medication and/or dosage during the study period.
* If female of childbearing potential, has a negative urine pregnancy test at Visit 1 and uses, or agrees to use, for the duration of the study, a medically acceptable form of contraception as determined by the investigator.
* Complete abstinence from intercourse from 2 weeks prior to administration of study drug throughout the study, and for a time interval after completion or premature discontinuation from the study to account for elimination of the study drug (a minimum of 7 days); or,
* Surgically sterile (hysterectomy or tubal ligation or otherwise incapable of pregnancy); or,
* Sterilization of male partner; or,
* Intrauterine device with published data showing lowest expected failure rate is less than 1% per year; or,
* Double barrier method (i.e., 2 physical barriers OR 1 physical barrier plus spermicide) for a least 1 month prior to Visit 1 and throughout study; or,
* Hormonal contraceptives for at least 3 months prior to Visit 1 and throughout study.

Exclusion Criteria:

Subject

* Is unable to understand the study requirements, the informed consent, or complete headache records as required per protocol.
* Is pregnant, actively trying to become pregnant, or breast-feeding.
* Has experienced the following migraine variants: basilar migraine, aura without headache, familial hemiplegic migraine, complicated migraine, ophthalmoplegic migraine and retinal migraine.
* Has a history of Medication Overuse Headache in the 3 months prior to study enrollment or during the Baseline Period.
* Has abused, in the opinion of the Investigator, any of the following drugs, currently or within the past 1 year: opioids, alcohol, barbiturates, benzodiazepine, cocaine
* Has an unstable neurological condition or a significantly abnormal neurological examination with focal signs or signs of increased intracranial pressure.
* Suffers from cardiovascular disease (ischemic heart disease, including angina pectoris, myocardial infarction, documented silent ischemia, or with Prinzmetal's angina); has symptoms of ischemic heart disease; have uncontrolled hypertension; has electrocardiogram (ECG) results outside normal limits for clinically stable patients as judged by the investigator.
* Has a history of asthma, allergy, or nasal polyps developing for the first time over the age of 40.
* Has a history of peptic ulcer disease requiring therapeutic intervention in the year prior to study enrollment.
* Has a history of bleeding peptic ulcer disease or perforation of the stomach or intestine.
* Has a history of bleeding disorder.
* Has history of Non-steroidal anti-inflammatory drug (NSAID) induced gastritis, esophagitis, or duodenitis.
* Suffers from a serious illness, or an unstable medical condition that could require hospitalization, or could increase the risk of adverse events.
* Has significant (as determined by the investigator) cardiovascular risk factors that may include uncontrolled high blood pressure, post-menopausal women, males over 40 years old, hypercholesterolemia, obesity, diabetes mellitus, smoking, or a family history of cardiovascular disease in a 1st degree relative.
* Has a psychiatric condition, in the opinion of the investigator that may affect the interpretation of efficacy and safety data or contraindicates the subject's participation in the study.
* Has hypersensitivity, intolerance, or contraindication to the use of sumatriptan, any of its components, or any other 5-hydroxytryptamine1 (5-HT1) agonist.
* Has a hypersensitivity, intolerance, or contraindication to the use of naproxen, any of its components, or any other non-steroidal anti-inflammatory drug including aspirin and cyclooxygenase-2 (COX-2) inhibiting agents.
* Is currently taking a migraine prophylactic medication containing an ergotamine or ergot derivative such as dihydroergotamine (DHE) or methysergide.
* Has taken, or plans to take, a monoamine oxidase inhibitor (MAOI) including herbal preparations containing St. John's wort (Hypericum perforatum), anytime within the 2 weeks prior to screening through 2 weeks post final study treatment.
* Has received any investigational agents within 30 days prior to Visit 1.
* Plans to participate in another clinical study at any time during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-09; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Cady, MD, Principal Investigator — Clinvest
Locations (2):
- United States (2):
  - Clinvest, Springfield, Missouri
  - Texas Headache Associates, San Antonio, Texas

REFERENCES:
- [Derived] Cady R, Nett R, Dexter K, Freitag F, Beach ME, Manley HR. Treatment of chronic migraine: a 3-month comparator study of naproxen sodium vs SumaRT/Nap. Headache. 2014 Jan;54(1):80-93. doi: 10.1111/head.12210. Epub 2013 Sep 10. PMID 24020994

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from date of Institutional Review Board (IRB) approval (8-3-10) until date last patient enrolled (1-30-12). Subjects were recruited from general population at two clinical research centers.
Pre-assignment Details: Subjects completed a 30 day Baseline period between Visit 1 and Visit 2 before Randomization. Subjects must have had 15 or more headache days during the 30 day Baseline period in order to be randomized into the study Treatment periods. Fifty-six subjects were screened for study, however only 28 subjects randomized for treatment due to screen fail.
Groups:
- Sumatriptan/Naproxen Sodium: In Treatment Period Month 1: Subjects randomized to Sumatriptan/Naproxen Sodium will treat daily with 1 tablet Sumatriptan/Naproxen Sodium (sumatriptan 85mg / naproxen sodium 500mg) per day x 30 days. Subjects will be provided with 30 tablets of Sumatriptan/Naproxen Sodium for rescue. In Treatment Period Months 2 and 3: Subjects randomized to Sumatriptan/Naproxen Sodium will be provided with 14 tablets of Sumatriptan/Naproxen Sodium to treat on 14 or fewer days per month. Subjects will be provided with 14 tablets of Sumatriptan/Naproxen Sodium per month for rescue.
Period: Overall Study
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Started | 16 | 12
Completed | 15 | 5
Not Completed | 1 | 7
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 1 | 5
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Sumatriptan/Naproxen Sodium: In Treatment Period Month 1: Subjects randomized to Treximet will treat daily with 1 tablet Treximet (sumatriptan 85mg / naproxen sodium 500mg) per day x 30 days. Subjects will be provided with 30 tablets of Treximet for rescue. In Treatment Period Months 2 and 3: Subjects randomized to Treximet will be provided with 14 tablets of Treximet to treat on 14 or fewer days per month. Subjects will be provided with 14 tablets of Treximet per month for rescue.
- Naproxen Sodium: In Treatment Period Month 1: Subjects randomized to naproxen will treat daily with 1 tablet naproxen 500mg per day x 30 days. Subjects will be provided with 30 tablets of naproxen 500mg for rescue. In Treatment Period Months 2 and 3: Subjects randomized to naproxen will be provided with 14 tablets of naproxen 500mg to treat on 14 or fewer days per month. Subjects will be provided with 14 tablets of naproxen 500mg per month for rescue.
- Total: Total of all reporting groups
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium | Total
Number analyzed (Participants) | 16 | 12 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 12 | 28
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.8 (12.6) | 37.0 (8.6) | 40.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 16 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of Migraine Headache Days Compared to Baseline
Description: Comparing the number of migraine headache days during Baseline Period days 1-30 to number of migraine headache days reported in Treatment Period days 91-120 in the Sumatriptan/Naproxen Sodium arm versus (vs.) Naproxen Sodium arm. Percent change=[(total headache days during Treatment Period Month 3(days 91-120)-total headache days during Baseline(days 1-30)/total headache days during Baseline(days 1-30)]*100%)
Time Frame: Day 121 (following 30 day Baseline Period and Treatment Period days 91-120.
Measure: Mean (Standard Deviation); unit: percent migraine headache days per month
Groups:
- Sumatriptan/Naproxen Sodium: In Treatment Period Month 1: Subjects randomized to Sumatriptan/Naproxen will treat daily with 1 tablet Sumatriptan/Naproxen per day x 30 days. Subjects will be provided with 30 tablets of Sumatriptan/Naproxen for rescue. In Treatment Period Months 2 and 3: Subjects randomized to Sumatriptan/Naproxen will be provided with 14 tablets of Sumatriptan/Naproxen to treat on 14 or fewer days per month. Subjects will be provided with 14 tablets of Sumatriptan/Naproxen per month for rescue.
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 15 | 5
percent migraine headache days per month | -8.06 (32.9) | -56.37 (36.2)

2. Secondary Outcome: Percent Change of Migraine Headache Days in All Treatment Periods Compared to Baseline
Description: Comparing number of migraine headache days from Baseline to Treatment Period Months 1, 2, and 3 in the Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm.
  Comparing the number of migraine headache days reported from Baseline Period days 1-30 to number of migraine headache days reported in Treatment Period days Months 1(days 31-60), 2(days 61-90),and 3(days 91-120)in the Sumatriptan/Naproxen Sodium arm versus (vs.) Naproxen Sodium arm. Each treatment period month percent change was individually compared to Baseline. The following formula was used for each treatment period calculation.
  e.g. percent change=[(total headache days during Treatment Period Month 3(days 91-120)-total headache days during Baseline(days 1-30)/total headache days during Baseline(days 1-30)]*100%)
Time Frame: Baseline Period (days 1-30) collected at Day 31, Treatment Period Months 1, 2, and 3 collected at Days 61, 91, and 121, respectively.
Measure: Mean (Standard Deviation); unit: percent migraine headache days per month
Groups:
- Sumatriptan/Naproxen Sodium: In Treatment Period Month 1: Subjects randomized to Sumatriptan/Naproxen Sodium will treat daily with 1 tablet Sumatriptan/Naproxen Sodium per day x 30 days. Subjects will be provided with 30 tablets of Sumatriptan/Naproxen Sodium for rescue. In Treatment Period Months 2 and 3: Subjects randomized to Sumatriptan/Naproxen Sodium will be provided with 14 tablets of Sumatriptan/Naproxen Sodium to treat on 14 or fewer days per month. Subjects will be provided with 14 tablets of Sumatriptan/Naproxen Sodium per month for rescue.
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 15 | 5
percent migraine headache days per month
  Baseline to Treatment Period Month 1 | -26.22 (31.4) | -61.55 (23.9)
  Baseline to Treatment Period Month 2 | -2.96 (23.7) | -45.42 (36.0)
  Baseline to Treatment Period Month 3 | -8.06 (32.9) | -56.37 (36.2)

3. Secondary Outcome: Migraine Headache Duration From Onset to Pain Free
Description: Comparing mean migraine duration from onset to pain free from Baseline Period (Days 1-30), to each of the Treatment Period Months 1(days 31-60), 2(days 61-90), and 3(days 91-120) in Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm. Percent change was calculated by determining percent change in each subject, from each Treatment Period month compared to Baseline. The following formula was used for each treatment period month calculation.
  e.g. Percent change=[(mean migraine duration from onset to pain free during Treatment Period Month 3(days 91-120)-mean migraine duration from onset to pain free during Baseline(days 1-30)/mean duration from onset to pain free during Baseline(days 1-30)]*100%)
Time Frame: Baseline Period collected at Day 31, Treatment Period Months 1, 2, and 3 collected at Days 61, 91, and 121 respectively.
Measure: Mean (Standard Deviation); unit: percent hours of migraine duration
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 15 | 5
percent hours of migraine duration
  Baseline to Treatment Period Month 1 | 167.83 (230.48) | 26.37 (13.11)
  Baseline to Treatment Period Month 2 | 176.18 (227.97) | 28.91 (21.21)
  Baseline to Treatment Period Month 3 | 151.49 (224.53) | 19.65 (30.82)

4. Secondary Outcome: Migraine Headache Duration From Time of Treatment to Pain Free
Description: Comparing mean migraine duration from time of treatment to pain free from Baseline Period (Days 1-30), to each of the Treatment Period Months 1(days 31-60), 2(days 61-90), and 3(days 91-120) in Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm. Percent change was calculated by determining percent change in each subject, from each Treatment Period month compared to Baseline. The following formula was used for each treatment period month calculation.
  e.g. Percent change=[(mean migraine duration from time of treatment to pain free during Treatment Period Month 3(days 91-120)-mean migraine duration from time of treatment to pain free during Baseline(days 1-30)/mean duration from time of treatment to pain free during Baseline(days 1-30)]*100%)
Time Frame: Baseline Period collected at Day 31, Treatment Period Months 1, 2, and 3 collected at Days 61, 91, and 121 respectively.
Measure: Mean (Standard Deviation); unit: percent hours of migraine duration
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 15 | 5
percent hours of migraine duration
  Baseline to Treatment Period Month 1 | 176.70 (233.18) | 24.58 (12.21)
  Baseline to Treatment Period Month 2 | 175.78 (228.08) | 28.45 (21.03)
  Baseline to Treatment Period Month 3 | 151.12 (224.45) | 23.15 (38.78)

5. Secondary Outcome: Migraine Headache Days With Greater Than 50% Reduction
Description: Number of subjects with at least 50% reduction in number of migraine headache days reported in Baseline vs. Treatment Period months 1(days 31-60), 2(days 61-90), and 3(days 91-120)in the Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm.
Time Frame: Baseline Period collected at Day 31, Treatment Period Months 1, 2, and 3 collected at Days 61, 92, and 121 respectively.
Measure: Number; unit: participants
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 15 | 5
participants
  Baseline to Treatment Period Month 1 | 3 | 4
  Baseline to Treatment Period Month 2 | 0 | 3
  Baseline to Treatment Period Month 3 | 3 | 4

6. Secondary Outcome: Percent Change of Doses of Study Medication
Description: Comparing the number of doses of study medication taken during Baseline Period(days 1-30) of triptans(Group A) and non-steroidal anti-inflammatory drugs(NSAIDS)(Group B)to the number of doses of study medication taken during Treatment Period Months 1(days 31-60), 2(days 61-90), and 3(days 91-120)in the Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm.
  e.g.Percent change=[(number of doses of study medication during Treatment Period Month 3(days 91-120)-number of doses of study medication during Baseline(days 1-30)/number of doses of study medication during Baseline(days 1-30)]*100%).
Time Frame: Baseline Period collected at Day 31, Treatment Period Months 1, 2, and 3 collected at Days 61, 92, and 121 respectively.
Measure: Mean (Standard Deviation); unit: percent doses of study medication
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 15 | 5
percent doses of study medication
  Baseline to Treatment Period Month 1 | 173.8 (194) | 825.6 (1649.9)
  Baseline to Treatment Period Month 2 | 40.1 (84) | 239.8 (575.8)
  Baseline to Treatment Period Month 3 | 40.0 (147) | 135.6 (379.33)

7. Secondary Outcome: Migraine Disability Assessment(MIDAS)Questionnaire Total Score
Description: Change in Migraine Disability Assessment (MIDAS) total score (effect migraine headaches have on subjects daily function) from Baseline (Day 31) to 3 months after Baseline to end of Treatment Period Month 3(Day 121) following final dose of study medication in the Sumatriptan/Naproxen Sodium arm vs. the Naproxen Sodium arm.
  Total score of disability ranges:
  * 0 to 5, MIDAS Grade I, Little or no disability
  * 6 to 10, MIDAS Grade II, Mild disability
  * 11 to 20, MIDAS Grade III, Moderate disability
  * 21+, MIDAS Grade IV, Severe disability Score ranges from 0-450. No subscales are present.
Time Frame: Baseline MIDAS collected at Day 31, Post final dose study at Day 121.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Sumatriptan/Naproxen Sodium: In Treatment Period Month 1: Subjects randomized to Sumatriptan/Naproxen Sodium will treat daily with 1 tablet Sumatriptan/Naproxen Sodium (sumatriptan 85 mg / naproxen sodium 500 mg) per day x 30 days. Subjects will be provided with 30 tablets of Sumatriptan/Naproxen Sodium for rescue. In Treatment Period Months 2 and 3: Subjects randomized to Sumatriptan/Naproxen Sodium will be provided with 14 tablets of Sumatriptan/Naproxen Sodium to treat on 14 or fewer days per month. Subjects will be provided with 14 tablets of Sumatriptan/Naproxen Sodium per month for rescue.
- Naproxen Sodium: In Treatment Period Month 1: Subjects randomized to Naproxen Sodium will treat daily with 1 tablet Naproxen Sodium 500 mg per day x 30 days. Subjects will be provided with 30 tablets of Naproxen Sodium for rescue. In Treatment Period Months 2 and 3: Subjects randomized to Naproxen Sodium will be provided with 14 tablets of Naproxen Sodium to treat on 14 or fewer days per month. Subjects will be provided with 14 tablets of Naproxen Sodium per month for rescue.
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 15 | 5
scores on a scale
  Day 31 | 76.6 (38.6) | 81.2 (52.9)
  Day 121 | 56.3 (44.5) | 16.4 (9.2)

8. Secondary Outcome: Compliance With Lifestyle Changes
Description: Self-assessed grade of compliance with lifestyle modification changes (where A=1, B=2, C=3, D=4, and F=5) in the Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm. Lower scores indicate a better outcome. Higher scores indicate a worse outcome.
Time Frame: Day 121
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 15 | 5
Units on a scale | 2.00 (0.65) | 2.40 (0.55)

ADVERSE EVENTS:
Groups:
- Naproxen Sodium: In Treatment Period Month 1: Subjects randomized to Naproxen Sodium will treat daily with 1 tablet Naproxen Sodium per day x 30 days. Subjects will be provided with 30 tablets of Naproxen Sodium for rescue. In Treatment Period Months 2 and 3: Subjects randomized to Naproxen Sodium will be provided with 14 tablets of naproxen 500mg to treat on 14 or fewer days per month. Subjects will be provided with 14 tablets of Naproxen Sodium per month for rescue.
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Serious Adverse Events (participants affected / at risk) | 1/16 | 1/12
Other Adverse Events (participants affected / at risk) | 9/16 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sumatriptan/Naproxen Sodium (N=16) | Naproxen Sodium (N=12)
Cholecystitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Menorragia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sumatriptan/Naproxen Sodium (N=16) | Naproxen Sodium (N=12)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Common Cold (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 1 (1) | 1 (1)
Elevated Blood Pressure (Cardiac disorders) | 1 (1) | 0 (0)
Enhanced Smell (General disorders) | 0 (0) | 1 (1)
Fever (Infections and infestations) | 1 (1) | 1 (1)
Flu (Infections and infestations) | 1 (1) | 1 (1)
Fluid in Ears (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (4)
Nausea with Fatty Foods (Gastrointestinal disorders) | 1 (1) | 0 (0)
Numb Feeling in Head (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain Behind Eyes (General disorders) | 0 (0) | 1 (1)
Right Ankle Sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right Leg Ulcer (Infections and infestations) | 1 (1) | 0 (0)
Sinus Burning Sensation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Infection (Infections and infestations) | 0 (0) | 1 (1)
Sore Throat (General disorders) | 1 (1) | 0 (0)
Stomach Burn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Strep Throat (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Worsening Stress (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less